CLINICAL TRIAL: NCT06700564
Title: The Diagnostic Efficacy and Lesion Detection Advantages of 18F-FDG PET/CT and Enhanced MRI in Hepatic Malignancies
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024212
Record Dates: First submitted 2024-10-22; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Hepatoma
Keywords: Hepatoma; pet/mr; contrast-enhanced MR
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- research group: This study adopts a prospective research design, with 60 patients suspected of having liver mass undergoing 18F-FDG PET/enhanced MR examination over one year. The inclusion criteria are as follows: age ≥ 18 years old; Patients suspected of having liver metastasis or liver lesions, based on clinical symptoms and laboratory tests (such as alpha-fetoprotein level); Preliminary findings from other routine imaging examinations; Able to perform 18F-FDG PET/MR examination and agree to follow the research procedure. The exclusion criteria are as follows: patients with a history of allergy to MR contrast agents; Pregnant or lactating women; Patients with severe heart disease, renal failure, liver failure, etc; Patients who are unable to cooperate in completing PET/MR examinations. This study passed the ethical review of Shanghai Oriental Hospital, and patients signed informed consent forms after enrollment.
  Interventions: Other: PET scan of FDG

INTERVENTIONS:
Other: PET scan of FDG — The enrolled patients will undergo PET examination, and the radiation dose generated during the examination will not cause physiological damage to the patients

SUMMARY:
Liver disease is a major challenge for global public health, covering a wide range from mild liver dysfunction to serious diseases such as cirrhosis and liver cancer. Globally, the high incidence rate and mortality of liver diseases have led to a huge socio-economic burden, especially in developing countries. Primary liver cancer, especially hepatocellular carcinoma (HCC), is the fifth most common cancer and the third leading cause of cancer death worldwide. In addition, the liver is a common site of metastasis for various cancers, and the occurrence of liver metastasis significantly affects the prognosis and treatment strategies of patients. In this context, accurately diagnosing the nature of liver lesions has become the key to improving patient treatment outcomes. Distinguishing between benign and malignant liver lesions is crucial for avoiding unnecessary invasive interventions and ensuring timely and appropriate treatment. Similarly, timely identification of liver metastases is crucial for the overall management and improvement of survival rates in cancer patients.

Traditional imaging techniques such as ultrasound, computed tomography (CT), and magnetic resonance imaging (MRI) have been widely used for the detection and characterization of liver lesions, but they have limitations in diagnostic specificity and sensitivity, limited recognition of specific pathological features, and insufficient ability to detect small metastases. Positron emission tomography/computed tomography (PET/CT), as a widely used fusion imaging technique, combines the metabolic information of PET with the anatomical information of CT, demonstrating unique value in the diagnosis and treatment evaluation of various tumors. However, PET/CT has specific limitations in its application in liver diseases, especially in analyzing small liver lesions and distinguishing between benign and malignant tumors in the context of cirrhosis, which may be challenging. In addition, the radiation exposure caused by CT components is a significant issue that cannot be ignored in PET/CT examinations.

Relatively speaking, PET/MR combined with 18F-fluorodeoxyglucose (18F-FDG)provides a new diagnostic possibility, especially when used in conjunction with abdominal-enhanced MR on the same machine, which is expected to further improve diagnostic accuracy. However, despite the theoretical superiority of this technology over traditional methods, the actual degree of improvement, scope of application, and impact on clinical decision-making are still unclear. Therefore, despite high expectations for this technology, it is necessary to conduct a comprehensive study to evaluate the specific benefits of 18F-FDG PET/MR combined with abdominal-enhanced MR in the diagnosis of liver lesions, the particular degree of improvement in diagnostic accuracy, and its potential contribution to improving patient treatment outcomes. This not only helps to validate the practical application value of this technology in the diagnosis of liver lesions but also provides evidence for clinical doctors to optimize and personalize patient diagnosis and treatment plans. The results of this study will provide the scientific basis for future clinical practice, ensuring the effective and cost-effective application of this technology in the management of liver diseases.

DETAILED DESCRIPTION:
This study is a prospective research design, enrolling 60 patients with suspected liver masses over a one-year period, who will undergo 18F-FDG PET/CT and enhanced MRI examinations.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old; Preliminary findings from other routine imaging examinations;
2. Patients suspected of having liver metastasis or liver lesions, based on clinical symptoms and laboratory tests (such as alpha-fetoprotein levels);
3. Preliminary findings from other routine imaging examinations;
4. Able to perform 18F-FDG PET/MR examination and agree to follow the research procedure.

Exclusion Criteria:

1. Patients with a history of allergy to MR contrast agents;
2. Pregnant or lactating women;
3. Patients with severe heart disease, renal failure, liver failure, etc;
4. Patients who are unable to cooperate in completing PET/MR examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with hepatocellular cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Radioactive uptake | After the patient signs the informed consent form and completes the scan, an average of 2 days.
  Assess the glucose uptake of the lesions.
manifestations of lesions on MR | After the patient signs the informed consent form and completes the scan, an average of 2 days.
  Two physicians will collaboratively document the dimensions of liver lesions.
manifestations of lesions on MR | After the patient signs the informed consent form and completes the scan, an average of 2 days.
  Two physicians will collaboratively assess the quantity of lesions.
Signal characteristics on MRI | After the patient signs the informed consent form and completes the scan, an average of 2 days.
  Evaluating the MR features of liver lesions, including T1 weighted, T2 weighted, diffusion-weighted imaging (DWI) characteristics, and enhanced features.

IPD SHARING:
Plan to Share IPD: No
In order to better protect patient privacy, the trial data will not be made public. Researchers can contact us via email to obtain the data.